CLINICAL TRIAL: NCT00480558
Title: A Phase I Study Evaluating the Safety and Immunogenicity of a New TB Vaccine, MVA85A, in Asymptomatic Volunteers Who Are Infected With Either Mycobacterium Tuberculosis (M.tb.), Human Immunodeficiency Virus (HIV) or Both
Brief Title: A Study of MVA85A, in Asymptomatic Volunteers Infected With TB, HIV or Both
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB011
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: HIV Infections; TB
Keywords: HIV; MVA85A; TB; Tuberculosis; Human Immunodeficiency Virus; Safety; Immunogenicity; Efficacy; Treatment Naive
MeSH Terms: conditions — HIV Infections; Tuberculosis; Acquired Immunodeficiency Syndrome | interventions — MVA 85A; MVA Pfs25-IMX313 malaria vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Group 1: M. tb
  Interventions: Biological: MVA 85A
- 2 (Active Comparator): Group 2: HIV (not on antiretrovirals [ARV])
  Interventions: Biological: MVA 85A
- 3 (Active Comparator): Group 3: M. tb and HIV (not on ARV)
  Interventions: Biological: MVA 85A
- 4 (Active Comparator): Group 4: M. tb and HIV (on ARV)
  Interventions: Biological: MVA 85A

INTERVENTIONS:
Biological: MVA 85A — Modified vaccinia Ankara virus expressing antigen 85A from M. tuberculosis. Dose is 5x10^7
  Other Names: TB Vaccine; modified vaccinia virus Ankara

SUMMARY:
This study is designed to evaluate the safety of MVA85A in asymptomatic volunteers in South Africa who are infected with M.tb, HIV or both. A single vaccination with MVA85A, when administered at a dose of 5 x 107pfu intradermally, is safe and highly immunogenic in mycobacterially naïve individuals, BCG vaccinated individuals and M.tb latently infected individuals. We will use the same vaccination regime in this study. Participants will be defined as being infected with M.tb.if they have a positive Elispot response to ESAT6 or CFP10. Participants will be defined as being infected with HIV.if they have a positive HIV rapid test (Determine®, Abbott Laboratories) followed by a positive HIV ELISA result. Participants will be identified from the general population living in Worcester, Western Cape, South Africa

DETAILED DESCRIPTION:
Prime-boost immunization strategies Heterologous prime-boost immunization strategies involve giving two different vaccines, each encoding the same antigen, several weeks apart. Using a DNA prime-recombinant modified vaccinia virus Ankara (MVA) boost induces higher levels of antigen specific CD4+ and CD8+ T cells than using homologous boosting with the same vector in a number of different disease models (Schneider, 1998; McShane, 2001). Given the protective efficacy of BCG in childhood, ideally BCG would be the priming immunization in such a prime-boost strategy. In order to do this, we have focused on antigen 85A as a candidate antigen. Antigen 85A is highly conserved amongst all mycobacterial species and is present in all strains of BCG. Antigen 85A is a major secreted antigen from M. tuberculosis which forms part of the antigen 85 complex (A, B and C). This complex constitutes a major portion of the secreted proteins of both M.tb and BCG. It is involved in fibronectin binding within the cell wall and has mycolyltransferase activity. Antigen 85A is immunodominant in murine and human studies and is protective in small animals (Huygen, 1996).

Recombinant modified vaccinia virus Ankara (rMVA). Many viruses have been investigated as potential recombinant vaccines. The successful worldwide eradication of smallpox via vaccination with live vaccinia virus highlighted vaccinia as a candidate for recombinant use. The recognition in recent years that non- replicating strains of poxvirus such as MVA and avipox vectors can be more immunogenic than traditional replicating vaccinia strains has enhanced the attractiveness of this approach. MVA (modified vaccinia virus Ankara) is a strain of vaccinia virus which has been passaged more than 570 times though avian cells, is replication incompetent in human cell lines and has a good safety record. It has been administered to more than 120,000 vaccinees as part of the smallpox eradication programme, with no adverse effects, despite the deliberate vaccination of high risk groups (Stickl, 1974; Mahnel, 1994). This safety in man is consistent with the avirulence of MVA in animal models. MVA has six major genomic deletions compared to the parental genome severely compromising its ability to replicate in mammalian cells (Meher, 1991). No replication has been documented in non- transformed mammalian cells. Viral replication is blocked late during infection of cells but importantly viral and recombinant protein synthesis is unimpaired even during this abortive infection. The viral genome has been proven to be stable through a large series of passages in chicken embryo fibroblasts. Replication-deficient recombinant MVA has been seen as an exceptionally safe viral vector. When tested in animal model studies recombinant MVA's have been shown to be avirulent, yet protectively immunogenic as vaccines against viral diseases and cancer. Recent studies in severely immunosuppressed macaques have supported the view that MVA should be safe in immunocompromised humans (Akira, 2001; Stittelaar, 2001).

Safety of rMVAs in immunosuppression. There is now considerable preclinical and clinical data demonstrating the safety and immunogenicity of MVA as a viral vector in immunosuppression and HIV infection. Recombinant MVAs expressing HIV antigens have been administered to immunosuppressed macaques with no serious adverse events (Stittelaar et al, 2001). In addition, the safety of recombinant MVAs expressing HIV antigens and epitopes have now been evaluated in several Phase I clinical trials of HIV-infected subjects, both on and off antiretroviral therapy, with no serious adverse events (Cosma et al, 2003; Harrer et al 2005).

Preclinical data supporting this BCG prime-MVA85A boost strategy In BALB/c mice, using BCG as the priming immunization and then boosting with MVA85A induces higher levels of both antigen specific IFN-γ secreting CD4+ and CD8+ T cells and significantly greater levels of protection against aerosol challenge than after BCG alone (Goonetilleke et al, 2003). This regime has now been further evaluated in the more sensitive guinea pig aerosol challenge model with very encouraging results. Guinea pigs vaccinated with BCG and boosted with MVA85A, and then further boosted with a second recombinant viral vector expressing antigen 85A, fowlpox-85A (FP85A) showed significantly greater protection against challenge than guinea pigs vaccinated with BCG alone (Williams et al, 2005). This regime is also immunogenic in rhesus macaques, and protective (Verrek, personal communication).

Clinical data to date with MVA85A UK studies Over the last 3 years HM has established a clinical trial programme to evaluate the safety and immunogenicity of this BCG prime-MVA85A boost vaccination strategy in a series of Phase I studies. MVA85A was the first candidate TB vaccine to enter clinical trials anywhere in the world in September 2002, and is currently the only one in clinical trials in Africa. The design of these Phase I studies with MVA85A allowed for sequential vaccination of volunteer groups with a step-wise increase in mycobacterial exposure, to minimize the possibility of a Koch reaction. Trials were also conducted sequentially in the UK and The Gambia, as there is a greater degree of exposure to both environmental mycobacteria and M.tb in The Gambia. A Koch reaction describes the development of immunopathology in a person or animal with tuberculosis, when an exaggerated immune response to M.tb is stimulated. It was described in patients with TB disease when Koch performed his original studies employing mycobacteria as a type of therapeutic vaccination. It has now been demonstrated in the mouse model of therapeutic vaccination27. Available animal data suggest that these reactions do not occur in mice latently infected with M.tb, suggesting that such reactions may correlate with high bacterial load and that the Koch phenomenon may not pose a problem for vaccination of asymptomatic albeit latently infected humans25.

In the UK, 14 mycobacterially and BCG naïve, asymptomatic volunteers were recruited. and vaccinated twice with 5 x 107pfu MVA85A, administered intradermally at 3 week intervals. In these studies, MVA85A was found to be safe and well tolerated. All subjects experienced some local side-effects (redness, itching etc) which lasted for 3-7 days after vaccination. Approximately one third of subjects experienced some transient systemic symptoms (myalgia, headache) for the first 12-24 hours after vaccination. All local and systemic side-effects spontaneously resolved. There were no serious or severe adverse events in any of these studies.

The main immunological outcome used in these ongoing clinical trials is the ex-vivo interferon-gamma (IFN-γ) Elispot assay, which was used to assess specific T cell responses to tuberculin PPD, purified antigen 85 complex and pools of overlapping 15mer peptides spanning the length of antigen 85A. A single vaccination with MVA85A induced remarkably high levels of specific effector T cell responses 1 week after vaccination (mean IFN-γ Elispot response to PPD was 460 spots per million PBMC).

Next, the safety of MVA85A in volunteers previously vaccinated with BCG was demonstrated in 17 volunteers. The safety profile of MVA85A in these 17 volunteers was the same as in the BCG naïve group. These 17 volunteers showed even higher peak levels of antigen specific T cells (mean response to PPD was 917 spots per million PBMC) 1 week post-vaccination than those immunized with MVA85A alone. Perhaps more importantly for the induction of T cell memory, volunteers who were previously BCG vaccinated maintained significantly higher levels of antigen specific T cells after MVA85A for up to 24 weeks after vaccination, when compared to those volunteers vaccinated with either BCG or MVA85A alone (McShane et al, 2004).

The next trial to be conducted in the UK looked at the boosting efficacy of MVA85A when administered one month after BCG vaccination. 10 healthy, BCG naïve volunteers were vaccinated with BCG and one month later were boosted with MVA85A. Comparable safety and boosting efficacy was seen to the previous trial where the interval between BCG and MVA85A was 0.5-37 years.

The current ongoing study in the UK is designed to assess the safety and immunogenicity of MVA85A in asymptomatic volunteers who are latently infected with M.tb. Latent infection with M.tb describes a state where an individual is presumed to have a very low level persistent bacterial infection with no clinical or radiological evidence of disease, and yet has a detectable immune response against M.tb. Latent infection in this study is defined using specific diagnostic tests based on antigens that are absent from BCG and most environmental mycobacteria such as ESAT 6 and CFP 10, allowing an accurate diagnosis of latent M.tb infection to be made. Subjects for this study were recruited from TB contact clinics and vaccinated with a single dose of MVA85A. Follow-up involved detailed radiological and clinical assessment of the safety of this vaccine in this group. To date, 11 subjects have been vaccinated with MVA85A in this study and the safety and immunogenicity profile of MVA85A is identical to that seen in previous studies. Importantly there has been no clinical, radiological or immunological evidence of a Koch reaction. The Elispot responses to PPD, ESAT 6, CFP10, antigen 85A and other mycobacterial antigens are being monitored for 12 months following vaccination.

Gambian studies Following the success of the trials with MVA85A in the UK, a collaboration with the MRC unit in The Gambia was initiated. MVA85A was first evaluated in Phase I clinical trials in BCG naïve subjects (n = 11) and subsequently in BCG primed subjects (n=10). In these studies the safety and immunogenicity profile is comparable to that seen in the UK studies. In both the UK and The Gambian studies, MVA85A induces 5-10 fold higher immune responses than any other recombinant MVA in clinical trials. The most likely explanation for this is that the volunteers have some weak pre-existing anti-mycobacterial immunity induced by exposure to environmental mycobacteria, and this is being boosted by vaccination with MVA85A. When MVA85A is administered to BCG naïve subjects in the Gambia, the magnitude and kinetics of response resemble the BCG primed group in the UK, a finding that is likely to represent a greater degree of environmental priming in tropical climates.

South African studies A Phase II study of the safety and immunogenicity of MVA85A in healthy, M.tb uninfected and HIV uninfected adults in Cape Town commenced in August 2005. The studies with MVA85A at this site have begun in adults, as a safety requirement despite the fact that we already have safety and immunogenicity data in adults from both the UK and the Gambian studies. The population in South Africa is very different from the UK and Gambian populations in terms of both host genetics and mycobacterial exposure. There is considerably more M.tb exposure in South Africa than in the Gambia and the exposure to environmental mycobacterial is believed to be lower in South Africa than the Gambia. The BCG literature demonstrates wide variation in efficacy across geographical areas and it was important to confirm our findings in adults in Cape Town before proceeding to a study in adolescents. We aim to vaccinate 24 adults in total. These studies commenced in August 2005, and to date, 14 volunteers have been vaccinated. Encouragingly, the safety and immunogenicity results so far are comparable with the previous studies in the UK and the Gambia.

ELIGIBILITY:
Inclusion Criteria:

For all groups:

* Asymptomatic adults aged 21 to 50 years
* Chest x-ray normal with no evidence of past/present TB infection or disease or any other clinically significant finding
* Resident in or near Worcester for the duration of the vaccination study
* Willingness to allow the investigators to discuss the volunteer's medical history with the
* volunteer's usual doctor or HIV physician
* Agreement to refrain from blood donation during the course of the study
* Willing and able to provide written informed consent
* Willingness to undergo an HIV test

For the M.Tb infected- and M.Tb/HIV coinfected- groups:

• Screening Elispot positive (more than 50 spots/million PBMC): for either the pool of ESAT6 peptides and/or the pool of CFP10 peptides and screening Elispot positive for PPD.

• Positive Mantoux test. (>10mm induration)

For the HIV infected and M.Tb/HIV coinfected groups:

* HIV antibody positive; diagnosed at least 3 months previously
* CD4 count >300; nadir CD4 not < 300

Exclusion Criteria:

For all groups:

* Any deviation from the normal range in biochemistry or haematology blood tests or in urine analysis that is considered to be clinically significant
* Any previous ARV therapy
* Prior receipt of a recombinant MVA or Fowlpox vaccine
* Use of any investigational or non-registered drug, live vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune modifying drugs within six months of vaccination. (For corticosteroids, this will mean prednisolone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Pregnant/lactating female and any female who is willing or intends to become pregnant during the study
* Any AIDS defining illness
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Seropositive for hepatitis B surface antigen (HBsAg) and or hepatitis C (antibodies to HCV)
* Presence of any underlying disease that compromises the diagnosis and evaluation of response to the vaccine (including evidence of cardiovascular disease, history of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ), history of insulin requiring diabetes mellitus, any ongoing chronic illness requiring ongoing specialist supervision (e.g., gastrointestinal), and chronic or active neurological disease)
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any history of anaphylaxis in reaction to vaccination
* PI assessment of lack of willingness to participate and comply with all requirements of the protocol
* Any other finding which in the opinion of the investigator would significantly increase the risk of having an adverse outcome from participating in this protocol

For the M.Tb infected group (but not the HIV infected and M.Tb/HIV coinfected groups):

* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection and asplenia

For the HIV infected and M.Tb/HIV coinfected groups (but not the M.Tb infected/HIV uninfected group)

* CD4 count now more than 300 and CD4 nadir not less than 300

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety of a single intradermal injection of 5 x 107p.f.u. MVA85A. | One year

SECONDARY OUTCOMES:
To assess the effect of a single vaccination with MVA85A in asymptomatic participants who are infected with M.Tb or HIV or both on the immune response, both to antigen 85A (the antigen in the vaccine) and to ESAT6/CFP10 antigens (M.tb specific). | One year

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- University Cape Town, Cape Town, South Africa

REFERENCES:
- [Background] McShane H, Pathan AA, Sander CR, Keating SM, Gilbert SC, Huygen K, Fletcher HA, Hill AV. Recombinant modified vaccinia virus Ankara expressing antigen 85A boosts BCG-primed and naturally acquired antimycobacterial immunity in humans. Nat Med. 2004 Nov;10(11):1240-4. doi: 10.1038/nm1128. Epub 2004 Oct 24. PMID 15502839
- [Background] Goonetilleke NP, McShane H, Hannan CM, Anderson RJ, Brookes RH, Hill AV. Enhanced immunogenicity and protective efficacy against Mycobacterium tuberculosis of bacille Calmette-Guerin vaccine using mucosal administration and boosting with a recombinant modified vaccinia virus Ankara. J Immunol. 2003 Aug 1;171(3):1602-9. doi: 10.4049/jimmunol.171.3.1602. PMID 12874255
- [Background] Bejon P, Peshu N, Gilbert SC, Lowe BS, Molyneux CS, Forsdyke J, Lang T, Hill AV, Marsh K. Safety profile of the viral vectors of attenuated fowlpox strain FP9 and modified vaccinia virus Ankara recombinant for either of 2 preerythrocytic malaria antigens, ME-TRAP or the circumsporozoite protein, in children and adults in Kenya. Clin Infect Dis. 2006 Apr 15;42(8):1102-10. doi: 10.1086/501459. Epub 2006 Mar 14. PMID 16575727
- [Background] Huygen K, Content J, Denis O, Montgomery DL, Yawman AM, Deck RR, DeWitt CM, Orme IM, Baldwin S, D'Souza C, Drowart A, Lozes E, Vandenbussche P, Van Vooren JP, Liu MA, Ulmer JB. Immunogenicity and protective efficacy of a tuberculosis DNA vaccine. Nat Med. 1996 Aug;2(8):893-8. doi: 10.1038/nm0896-893. PMID 8705859
- [Background] McShane H, Brookes R, Gilbert SC, Hill AV. Enhanced immunogenicity of CD4(+) t-cell responses and protective efficacy of a DNA-modified vaccinia virus Ankara prime-boost vaccination regimen for murine tuberculosis. Infect Immun. 2001 Feb;69(2):681-6. doi: 10.1128/IAI.69.2.681-686.2001. PMID 11159955
- [Background] Colditz GA, Brewer TF, Berkey CS, Wilson ME, Burdick E, Fineberg HV, Mosteller F. Efficacy of BCG vaccine in the prevention of tuberculosis. Meta-analysis of the published literature. JAMA. 1994 Mar 2;271(9):698-702. PMID 8309034
- [Derived] Tanner R, Kakalacheva K, Miller E, Pathan AA, Chalk R, Sander CR, Scriba T, Tameris M, Hawkridge T, Mahomed H, Hussey G, Hanekom W, Checkley A, McShane H, Fletcher HA. Serum indoleamine 2,3-dioxygenase activity is associated with reduced immunogenicity following vaccination with MVA85A. BMC Infect Dis. 2014 Dec 3;14:660. doi: 10.1186/s12879-014-0660-7. PMID 25466778
- [Derived] Scriba TJ, Tameris M, Smit E, van der Merwe L, Hughes EJ, Kadira B, Mauff K, Moyo S, Brittain N, Lawrie A, Mulenga H, de Kock M, Makhethe L, Janse van Rensburg E, Gelderbloem S, Veldsman A, Hatherill M, Geldenhuys H, Hill AV, Hawkridge A, Hussey GD, Hanekom WA, McShane H, Mahomed H. A phase IIa trial of the new tuberculosis vaccine, MVA85A, in HIV- and/or Mycobacterium tuberculosis-infected adults. Am J Respir Crit Care Med. 2012 Apr 1;185(7):769-78. doi: 10.1164/rccm.201108-1548OC. Epub 2012 Jan 26. PMID 22281831